CLINICAL TRIAL: NCT02205281
Title: Partners in Health: A Couples-based Approach to Obesity Prevention.
Acronym: PIH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: California Polytechnic State University-San Luis Obispo (Other)
Collaborators: Dignity Health- French Hospital Medical Center (Unknown)
Responsible Party: Principal Investigator, Suzanne Phelan, Associate Professor, California Polytechnic State University-San Luis Obispo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 72514
Record Dates: First submitted 2014-07-29; First posted 2014-07-31 (Estimated); Last update posted 2020-08-28 (Actual); Status verified 2020-08

CONDITIONS: Obesity
Keywords: Overweight; Obese; Pregnancy; Weight Gain; Weight Loss
MeSH Terms: conditions — Obesity; Overweight; Weight Gain; Weight Loss

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard Care (No Intervention)
- Lifestyle Intervention (Experimental)
  Interventions: Behavioral: Lifestyle Intervention

INTERVENTIONS:
Behavioral: Lifestyle Intervention — The intervention is a multi-component program designed to prevent excessive gestational weight gain in overweight and obese women and to promote weight loss in their non-pregnant overweight and obese partners through modifications of diet, exercise, and behavioral strategies during pregnancy.
  Arms: Lifestyle Intervention

SUMMARY:
The purpose of this pilot study is to test the feasibility of an innovative, couples based approach to weight management during pregnancy. The primary hypothesis is that a couples-based behavioral weight management program will reduce the rate of gestational weight gain compared to standard care.

ELIGIBILITY:
Inclusion Criteria:

Pregnant Women

* >18 years old
* 15-22 weeks gestation
* BMI >= 25
* cohabitating with partner for at least 3 months or recently married
* willing to consent

Non-pregnant Partner

* BMI >= 25
* cohabitating with partner for at least 3 months or recently married
* willing to consent

Exclusion Criteria:

* Untreated medical or psychological problem
* Inability to be physically active

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-06 (Actual); Primary Completion 2018-05 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
Gestational weight gain | 16 weeks gestation, 35 weeks gestation
  Rate of gestational weight gain will be computed as difference between weights measured at study entry and gestational week 35; this difference will be divided by the number of weeks of observation during pregnancy (i.e., weeks between study entry and final pregnancy assessment). If gestational week 35 is unavailable, most proximal clinic visit weight will be used.

SECONDARY OUTCOMES:
Partner's weight loss | study entry, when pregnant partner reaches 35 weeks gestation
  Weight lost by the non-pregnant partner during the study will be assessed by subtracting their weight at the 35 week gestation visit from their study entry weight.

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne Phelan, PhD, Principal Investigator — Cal Poly
Locations (1):
- Cal Poly, San Luis Obispo, California, United States